CLINICAL TRIAL: NCT07364344
Title: A Single-Center,Open-Label Clinical Study on the Safety and Preliminary Efficacy of Hibernation-Like Therapy (Chlorpromazine and Promethazine) in Patients With Acute Ischemic Stroke (AIS) Eligible for Reperfusion Therapy.
Brief Title: Safety and Preliminary Efficacy of Hibernation-Like Therapy (Chlorpromazine and Promethazine) in Patients With Acute Ischemic Stroke (AIS) Eligible for Reperfusion Therapy.
Acronym: CHILL-S
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHILL-S; 3500-123203 (Registry Identifier: Capital Medical University); IIT-2025-YW055-02 (Registry Identifier: Ethics Committee of Zhoukou Central Hospital)
Record Dates: First submitted 2026-01-04; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Chlorpromazine; Promethazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hibernation-Like Therapy (Chlorpromazine and Promethazine) (Experimental)
  Interventions: Drug: Hibernation-like Therapy (Chlorpromazine and Promethazine, C+P)

INTERVENTIONS:
Drug: Hibernation-like Therapy (Chlorpromazine and Promethazine, C+P) — The escalating doses are Chlorpromazine and Promethazine (C+P) at the following combinations: 50mg+50mg, 62.5mg+62.5mg, 75mg+75mg, and 100mg+100mg.Dose escalation will follow the "3+3" rule. Based on the dose-escalation results, dose expansion will be initiated at an appropriate time. The dose-expansion phase will consist of three cohorts: two cohorts receiving C+P and one cohort receiving an intravenous infusion of 50ml normal saline at room temperature (infusion rate also 50ml/h) prior to endovascular treatment. The two C+P dose groups for expansion will be selected based on the dose-escalation results. Patients will receive the study drug followed by reperfusion therapy. The administration method is the same as in the dose-escalation phase.

SUMMARY:
This is a single-center, dose-escalation and dose-expansion Phase I study designed to evaluate the safety of hibernation-like therapy (Chlorpromazine and Promethazine, C+P) and observe improvements in infarct volume in patients with AIS eligible for reperfusion therapy.

DETAILED DESCRIPTION:
Part A is the dose-escalation phase, and Part B is the dose-expansion phase. Both Part A and Part B will enroll subjects with AIS who are eligible for endovascular treatment based on multimodality imaging assessment and who meet all inclusion criteria and none of the exclusion criteria as evaluated by the investigator. Successfully screened patients will first enter the dose-escalation study. The escalating doses are Chlorpromazine and Promethazine (C+P) at the following combinations: 50mg+50mg, 62.5mg+62.5mg, 75mg+75mg, and 100mg+100mg.

Dose escalation will follow the "3+3" rule, with a planned enrollment of 12-24 subjects. Based on the dose-escalation results, dose expansion will be initiated at an appropriate time. The dose-expansion phase will consist of three cohorts: two cohorts receiving C+P and one cohort receiving an intravenous infusion of 50ml normal saline at room temperature (infusion rate also 50ml/h) prior to endovascular treatment. The two C+P dose groups for expansion will be selected based on the dose-escalation results. Patients will receive the study drug followed by reperfusion therapy. The administration method is the same as in the dose-escalation phase. The dose-expansion phase plans to enroll 33 subjects (10 subjects each in the two C+P cohorts and 13 subjects in the normal saline cohort). See the figure below for details.

C+P is administered intravenously. The administration regimen involves dissolving C+P in 50ml of normal saline at room temperature and infusing it intravenously at a rate of 50ml/h (complete infusion over 1 hour). Subsequently, the patient will undergo endovascular thrombectomy for recanalization.

The DLT observation period in the dose-escalation phase is 3 days after administration. Escalation to the next dose cohort may proceed only after the DLT observation period for the current cohort is completed and safety is confirmed.

Patients will receive only a single administration during both the dose-escalation and dose-expansion phases. Within 24 hours after completing endovascular thrombectomy, patients will undergo ECG monitoring with close observation of vital signs and changes in consciousness level. Vital signs will continue to be monitored for up to 72 hours post-thrombectomy, and imaging follow-up will be performed at 48 ±12 hours.

Study Objectives:

* Primary Objective: To evaluate the safety of hibernation-like therapy (Chlorpromazine + Promethazine, C+P) in patients with acute ischemic stroke (AIS) eligible for reperfusion therapy, to observe the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) across different C+P dose cohorts, and to determine the recommended phase 2 dose (RP2D).
* Secondary Objective: To evaluate the efficacy of hibernation-like therapy (C+P) in patients with AIS eligible for reperfusion therapy.
* Exploratory Objective: To observe changes in metabolomics at 3 hours post-administration compared to baseline.

Endpoints:

* Primary Endpoint: Observation of DLT and MTD across different C+P dose cohorts to determine the RP2D.
* Secondary Endpoints:

  * Improvement in cerebral infarct volume (mL) at 48 ±12 hours post-treatment compared to pre-treatment.
  * Improvement in the National Institutes of Health Stroke Scale (NIHSS) score at 24 hours post-treatment compared to baseline.
  * Assessment of other safety parameters.
* Exploratory Endpoint: Changes in metabolomics at 3 hours post-administration compared to pre-administration.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or their legal guardian voluntarily agrees to participate by providing written informed consent, and agrees to comply with the trial treatment plan and visit schedule.
2. Male or female, aged 18 to 80 years (inclusive).
3. Diagnosis of acute ischemic stroke eligible for endovascular therapy.
4. Clinical signs and symptoms consistent with acute anterior circulation ischemic stroke, with a National Institutes of Health Stroke Scale (NIHSS) score between 6 and 20 (inclusive).

   Note: The NIHSS score ranges from 0 to 42, with higher scores indicating more severe neurological deficits. Classification:
   * *0-1: Normal or near-normal.*
   * *1-4: Minor stroke.*
   * *5-15: Moderate stroke.*
   * *15-20: Moderate to severe stroke.*
   * *21-42: Severe stroke.*
5. Time from stroke onset to planned drug administration is within 24 hours.
6. Pre-stroke modified Rankin Scale (mRS) score of 0 or 1.
7. Expected survival greater than 90 days.
8. Imaging Inclusion Criteria:

   * Pre-procedural angiographic evaluation (NCCT + CTA + CTP / DSA) confirms a large vessel occlusion (internal carotid artery or M1 segment of middle cerebral artery) consistent with clinical symptoms.
   * Alberta Stroke Program Early CT Score (ASPECTS) ≥ 6.
   * Perfusion-core mismatch: Ischemic core volume 5-70 mL, with a mismatch ratio (volume of hypoperfused tissue / volume of ischemic core) ≥ 1.8 and a mismatch volume ≥ 15 mL.
9. Adequate organ function at screening, defined as:

   * Platelet count > 100 × 10⁹/L.
   * Liver and renal function: ALT/AST ≤ 2.5 × upper limit of normal (ULN); Total bilirubin ≤ 1.5 × ULN; Creatinine clearance (Ccr) > 60 mL/min.
10. Female subjects of childbearing potential must agree to use effective contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the study and for 6 months after study completion. A negative pregnancy test is required within 7 days prior to enrollment. All subjects (male or female) must employ adequate contraceptive measures throughout the treatment period and for 6 months thereafter. (A negative pregnancy test result is mandatory for women of childbearing potential before enrollment).

Exclusion Criteria:

1. Presence of pathological fever at screening: axillary temperature ≥ 37.3°C or tympanic membrane temperature ≥ 37.9°C.
2. Clinical presentation suggestive of intracranial parenchymal hemorrhage or subarachnoid hemorrhage (even with normal imaging findings).
3. Stroke onset accompanied by seizures at screening, precluding accurate NIHSS assessment.
4. Coma or psychiatric disorders at screening that interfere with neurological evaluation.
5. Conditions contraindicating phenothiazine use at screening, such as Parkinson's disease, parkinsonism, basal ganglia disorders, bone marrow suppression, glaucoma, epilepsy, history of neuroleptic malignant syndrome, or history of hypersensitivity to phenothiazines.
6. History of severe infusion reactions deemed ineligible for inclusion upon evaluation.
7. History of allergy or anaphylactic shock to iodinated contrast agents.
8. Major surgery within 4 weeks prior to drug administration.
9. Blood glucose <50 mg/dL (2.78 mmol/L) or >400 mg/dL (22.20 mmol/L) prior to drug administration (fingerstick glucose results acceptable).
10. History of deep vein thrombosis within 6 months prior to drug administration.
11. Previous endovascular thrombectomy performed less than 3 months prior.
12. Clinically significant active bleeding (e.g., gastrointestinal or other) within 30 days prior to drug administration; coagulation factor abnormalities or bleeding tendency (e.g., on anticoagulants with INR ≥3 or PT ≥3×ULN). However, subjects may be enrolled without awaiting coagulation results if the investigator deems no coagulation dysfunction. Active infection requiring systemic therapy within 2 weeks prior to drug administration (e.g., active tuberculosis).
13. Clinically significant cardiac disease at screening, including but not limited to:

    * Uncontrolled hypertension (SBP >180 mmHg or DBP >105 mmHg after standard treatment) or hypotension (SBP ≤100 mmHg after standard treatment).
    * Unstable angina, myocardial infarction, or coronary artery bypass graft/stent placement within 6 months prior to drug administration.
    * History of chronic heart failure (NYHA Class 3-4), or valvular heart disease, deemed ineligible by the investigator.
14. Severe arrhythmia requiring treatment or presence of QT interval prolongation at screening, deemed ineligible by the investigator.
15. Severe systemic disease at screening deemed ineligible by the investigator, including but not limited to: pulmonary embolism, pulmonary hypertension, severe COPD, active tuberculosis, severe pneumonia, pneumothorax, severe atelectasis, severe pulmonary fibrosis, bronchopulmonary dysplasia, unstable pleural effusion, acute respiratory distress syndrome, irregular breathing patterns or other severe pulmonary diseases; severe hepatic or renal insufficiency such as cirrhosis, hepatic encephalopathy, ascites, obstructive jaundice, renal failure, or uremia.
16. Pregnant or lactating women.
17. Participation in an interventional clinical trial involving investigational drugs or medical devices within 28 days prior to screening.
18. Subjects considered inappropriate for inclusion by the investigator.

Imaging Exclusion Criteria:

1. CTA+CTP/DSA demonstrates excessive vascular tortuosity that may impede delivery of interventional devices.
2. Suspected cerebral vasculitis based on history and NCCT+CTA+CTP/DSA findings.
3. Suspected aortic dissection based on history and NCCT+CTA+CTP/DSA findings.
4. NCCT+CTA+CTP/DSA confirms occlusion in multiple vascular territories (e.g., bilateral anterior circulation or anterior/posterior circulation, extracranial carotid with intracranial tandem lesions), or clinical evidence of bilateral or multifocal infarction.
5. NCCT+CTA+CTP/DSA confirms moyamoya disease or moyamoya syndrome.
6. NCCT+CTP confirms significant mass effect with midline shift.
7. NCCT (or MRI) confirms presence of an intracranial tumor (except small meningiomas).
8. NCCT confirms presence of intracranial hemorrhage.
9. CTA misdiagnosis of large vessel occlusion (internal carotid artery or MCA M1 segment) where DSA angiography reveals no culprit vessel occlusion.
10. CTA misdiagnosis of a single anterior circulation large vessel occlusion where DSA angiography reveals occlusion of multiple major arterial trunks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Observation of DLT and MTD across different C+P dose cohorts to determine the RP2D. | From the initiation of Hibernation-Like Therapy until 7 days after treatment.

SECONDARY OUTCOMES:
Change in cerebral infarct volume (mL) at 48 ±12 hours post-treatment compared to pre-treatment. | From the start of Hibernation-Like Therapy to 48±12 hours after treatment.
Change in the National Institutes of Health Stroke Scale (NIHSS) score at 24 hours post-treatment compared to baseline. | From the start of Hibernation-Like Therapy to 24 hours after treatment.
Magnitude of vital sign changes (absolute differences in temperature, BP, and respiration post-C+P vs. baseline). | From the initiation of Hibernation-Like Therapy until 7 days after treatment.

OTHER OUTCOMES:
Ratio of specific metabolite downregulation after 3 hours of C+P therapy versus baseline (serum enrichment analysis). | From the start of Hibernation-Like Therapy to 3 hours after treatment.

IPD SHARING:
Plan to Share IPD: No
The number of subjects in this study was relatively small, making it easy to be precisely located. They don't want their health data to be leaked.

REFERENCES:
- [Result] Baron JC. Protecting the ischaemic penumbra as an adjunct to thrombectomy for acute stroke. Nat Rev Neurol. 2018 Jun;14(6):325-337. doi: 10.1038/s41582-018-0002-2. PMID 29674752
- [Result] Al-Mufti F, Amuluru K, Roth W, Nuoman R, El-Ghanem M, Meyers PM. Cerebral Ischemic Reperfusion Injury Following Recanalization of Large Vessel Occlusions. Neurosurgery. 2018 Jun 1;82(6):781-789. doi: 10.1093/neuros/nyx341. PMID 28973661
- [Result] Fisher M, Saver JL. Future directions of acute ischaemic stroke therapy. Lancet Neurol. 2015 Jul;14(7):758-67. doi: 10.1016/S1474-4422(15)00054-X. PMID 26067128
- [Result] Andrews BJ, Herskowitz I. The yeast SWI4 protein contains a motif present in developmental regulators and is part of a complex involved in cell-cycle-dependent transcription. Nature. 1989 Dec 14;342(6251):830-3. doi: 10.1038/342830a0. PMID 2689885
- [Result] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Result] Seners P, Turc G, Maier B, Mas JL, Oppenheim C, Baron JC. Incidence and Predictors of Early Recanalization After Intravenous Thrombolysis: A Systematic Review and Meta-Analysis. Stroke. 2016 Sep;47(9):2409-12. doi: 10.1161/STROKEAHA.116.014181. Epub 2016 Jul 26. PMID 27462117
- [Result] Tilley BC, Lyden PD, Brott TG, Lu M, Levine SR, Welch KM. Total quality improvement method for reduction of delays between emergency department admission and treatment of acute ischemic stroke. The National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Arch Neurol. 1997 Dec;54(12):1466-74. doi: 10.1001/archneur.1997.00550240020008. PMID 9400355
- [Result] Horne JA. A review of the biological effects of total sleep deprivation in man. Biol Psychol. 1978 Sep;7(1-2):55-102. doi: 10.1016/0301-0511(78)90042-x. PMID 747719
- [Result] Zuerrer M, Martin E, Boltshauser E. MR imaging of intracranial hemorrhage in neonates and infants at 2.35 Tesla. Neuroradiology. 1991;33(3):223-9. doi: 10.1007/BF00588222. PMID 1881539
- [Result] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116